CLINICAL TRIAL: NCT02887287
Title: Efficacy of Exclusive Enteral Nutrition in Adult Active Crohn's Disease
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, committee of the Sixth Affiliated Hospital of Sun Yat-sen University, Sun Yat-sen University
Other Study IDs: E2016008
Record Dates: First submitted 2016-08-29; First posted 2016-09-02 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-08

CONDITIONS: Efficacy of Exclusive Enteral Nutrition in Adult Active Crohn's Disease With Complications or Failure of Medical Treatment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Drug: EEN

SUMMARY:
The study aimed to prove EEN is effective for inducing early clinical remission, mucosal healing, promoting fistula closure and reducing the size of abscess to adult CD patients. They plan to include about 50 patients and observe the effect of EEN.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Patients with CD was diagnosed clinically according to previously established international criteria [9]
* The diagnosis of stricture, fistula and abdominal abscess was confirmed by ultrasound, CT enterography (CTE), and endoscopy. The bowel stricture should mainly cause by inflammation but not fibrosis.

Exclusion Criteria:

* Patients do not macth the inclusion criteria and those who refuse to taking part in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The detailed inclusion criteria included: 1. >18 years old 2. Patients with CD was diagnosed clinically according to previously established international criteria [9] 3. The diagnosis of stricture, fistula and abdominal abscess was confirmed by ultrasound, CT enterography (CTE), and endoscopy. The bowel stricture should mainly cause by inflammation but not fibrosis. Intolerance or failure to steroids or IFX was judged by medical history 4. The disease was in an active period.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2013-07; Primary Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Clinical remission after 12 weeks EEN | July 2013 to October 2015

CONTACTS AND LOCATIONS:
Locations (1):
- The six affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Yang Q, Gao X, Chen H, Li M, Wu X, Zhi M, Lan P, Hu P. Efficacy of exclusive enteral nutrition in complicated Crohn's disease. Scand J Gastroenterol. 2017 Sep;52(9):995-1001. doi: 10.1080/00365521.2017.1335770. Epub 2017 Jun 9. PMID 28598298